CLINICAL TRIAL: NCT03094195
Title: A Double-blind, Placebo-controlled, Randomized Dose Ranging Trial to Determine the Safety and Efficacy of Three Dose Levels of EMA401 in Reducing 24-hour Average Pain Intensity Score in Patients With Post-herpetic Neuralgia
Brief Title: Dose Response Study of EMA401 in Patients With Post-herpetic Neuralgia (PHN)
Acronym: EMPHENE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to pre-clinical toxicity data that became available after start of trial
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEMA401A2201
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Results first posted 2020-05-14 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Post-herpetic Neuralgia
Keywords: post-herpetic neuralgia; neuropathic pain; angiotensin II type 2 receptor antagonist; dose ranging
MeSH Terms: conditions — Neuralgia, Postherpetic; Neuralgia | interventions — EMA400

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EMA401 25mg BID (Experimental): Ema401 25 mg was administered orally twice a day
  Interventions: Drug: EMA401
- EMA401 100mg BID (Experimental): Ema401 100 mg was administered orally twice a day
  Interventions: Drug: EMA401
- Placebo BID (Placebo Comparator): Matching placebo capsules administered orally twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EMA401 — EMA401
  Arms: EMA401 100mg BID; EMA401 25mg BID
Drug: Placebo — Placebo
  Arms: Placebo BID

SUMMARY:
This study was designed to characterize dose response, and evaluate safety and efficacy of three different doses of EMA401 compared to placebo in patients with post-herpetic neuralgia (PHN).

DETAILED DESCRIPTION:
This was an interventional, randomized, parallel, placebo-controlled, dose ranging, double-blind treatment study consisting of 3 periods i.e. Screening, Treatment, and Treatment withdrawal. The study was planned in two cohorts. The initial cohort had three treatment arms i.e. Placebo b.i.d., EMA401 25 mg b.i.d., or EMA401 100 mg b.i.d. Following an unblinded safety review by an independent DMC, the second cohort was to have been initiated with an additional treatment arm i.e. EMA401 300 mg b.i.d.. Due to the premature study termination, the second cohort was not initiated. At the end of treatment period the 25mg BID and 100mg BID arms were re-randomized (1:1) to the same treatment or placebo. Placebo arm stayed on placebo. The planned duration of treatment period was 12 weeks and 1 week of treatment withdrawal at the end of treatment period. The study was terminated early due to pre-clinical toxicity data that became available after start of trial. Novartis implemented a Urgent Safety Measure (USM) which instructed sites to discontinue study treatment immediately and to have all patients return for additional laboratory assessments (full hematology including coagulation and clinical chemistry panel). Safety data from the USM was presented as a separate outcome measure table and not included in the Adverse Event section.

ELIGIBILITY:
Inclusion Criteria:

* At the time of Screening, must have had documented diagnosis of PHN (ICD-10 code B02.29), defined as pain in the region of the rash persisting for more than 6 months after onset of herpes zoster rash.
* Assessed as suffering from moderate to severe neuropathic pain across the Screening epoch (NRS ≥ 4).
* Patients must have had documented past and/or ongoing inadequate treatment response (having insufficient pain relief with treatment or inability to tolerate) to at least 2 different prescribed therapies commonly used to treat and considered effective by the Investigator for the treatment of PHN.
* Patient must have been willing to complete daily eDiary

Exclusion Criteria:

* History or had current diagnosis of electrocardiogram (ECG) abnormalities indicating significant risk of safety for patients participating in the study
* Had a major depressive episode within 6 months prior to Screening and/or a history of diagnosed recurrent major depressive disorder according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) diagnostic criteria
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.
* Had evidence of significant renal insufficiency or pre-existing liver condition
* Had platelets ≤ 100 x 10^9/L, or neutrophil count < 1.2 x 10^9/L (or equivalent), hemoglobin ≤ 100 g/L for women or hemoglobin ≤ 110 g/L for men.
* Patients who had a known diagnosis of diabetes and are stable on medication with a hemoglobin A1c > 8%. Those who did not have a known diagnosis of diabetes with a hemoglobin A1c > 7%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (55):
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Austria (2):
  - Novartis Investigative Site, Klagenfurt
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Pellenberg, Belgium
- Canada (3):
  - Novartis Investigative Site, Ontario, CAN
  - Novartis Investigative Site, Lévis, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Czechia (4):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Choceň
  - Novartis Investigative Site, Plzen-Bory
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Odense C, Denmark
- France (4):
  - Novartis Investigative Site, Boulogne-Billancourt
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Lille Cédex
  - Novartis Investigative Site, Nice
- Germany (8):
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Haar
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Wiesbaden
- Hungary (3):
  - Novartis Investigative Site, Esztergom, HUN
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Szeged
- Novartis Investigative Site, Rome, Italy
- Japan (8):
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Kawaguchi, Saitama
  - Novartis Investigative Site, Shizuoka, Shizuoka
  - Novartis Investigative Site, Kasukabe-shi, Tokyo
  - Novartis Investigative Site, Setagaya Ku, Tokyo
  - Novartis Investigative Site, Ōita
- Novartis Investigative Site, Oslo, Norway
- Poland (2):
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Warsaw
- Portugal (5):
  - Novartis Investigative Site, Almada
  - Novartis Investigative Site, Aveiro
  - Novartis Investigative Site, Leiria
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Slovakia (4):
  - Novartis Investigative Site, Dubnica nad Váhom, SVK
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Spišská Nová Ves
- Novartis Investigative Site, Seongnam-si, Gyeonggi-do, South Korea
- Spain (2):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona
- Novartis Investigative Site, Tainan, Taiwan
- United Kingdom (3):
  - Novartis Investigative Site, Darlington, Durham
  - Novartis Investigative Site, London, GBR
  - Novartis Investigative Site, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Rice ASC, Dworkin RH, Finnerup NB, Attal N, Anand P, Freeman R, Piaia A, Callegari F, Doerr C, Mondal S, Narayanan N, Ecochard L, Flossbach Y, Pandhi S. Efficacy and safety of EMA401 in peripheral neuropathic pain: results of 2 randomised, double-blind, phase 2 studies in patients with postherpetic neuralgia and painful diabetic neuropathy. Pain. 2021 Oct 1;162(10):2578-2589. doi: 10.1097/j.pain.0000000000002252. PMID 33675631
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=623

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two hundred thirty patients were screened.
Groups:
- EMA401 25mg BID DB: Ema401 25 mg was administered orally twice a day during double blind (DB) treatment period
- EMA401 100mg BID DB: Ema401 100 mg was administered orally twice a day during double blind (DB) treatment period
- Placebo BID DB: Matching placebo capsules administered orally twice a day during double blind (DB) treatment period
- EMA401 25mg BID -> EMA401 25mg BID TW; EMA401 25mg BID -> Placebo BID TW: Participants on EMA401 25mg were randomized 1:1 to EMA401 25mg or placebo at end of treatment period (week 12)
- EMA401 100mg BID -> EMA401 100mg BID TW; EMA401 100mg BID -> Placebo BID TW: Participants on EMA401 100mg were randomized 1:1 to EMA401 100mg or placebo at end of treatment period (week 12)
- Placebo BID -> Placebo BID TW: Participants on placebo remained on placebo at end of treatment period (week 12)
Period: Double-Blind Treatment Period (DB)
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB | Placebo BID DB | EMA401 25mg BID -> EMA401 25mg BID TW | EMA401 25mg BID -> Placebo BID TW | EMA401 100mg BID -> EMA401 100mg BID TW | EMA401 100mg BID -> Placebo BID TW | Placebo BID -> Placebo BID TW
Started | 43 | 43 | 43 | 0 | 0 | 0 | 0 | 0
Completed (Study completers completed the treatment phase regardless of completion of study treatment.) | 28 | 30 | 29 | 0 | 0 | 0 | 0 | 0
Not Completed | 15 | 13 | 14 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 12 | 10 | 11 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Treatment Withdrawal Period (TW)
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB | Placebo BID DB | EMA401 25mg BID -> EMA401 25mg BID TW | EMA401 25mg BID -> Placebo BID TW | EMA401 100mg BID -> EMA401 100mg BID TW | EMA401 100mg BID -> Placebo BID TW | Placebo BID -> Placebo BID TW
Started | 0 | 0 | 0 | 13 | 13 | 15 | 13 | 26
Completed | 0 | 0 | 0 | 13 | 13 | 15 | 13 | 26
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB | Placebo BID DB | Total
Number analyzed (Participants) | 43 | 43 | 43 | 129
Age, Customized [Number; unit: participants]
  18 - 64 years | 4 | 8 | 7 | 19
  65 - 84 years | 36 | 34 | 36 | 106
  ≥ 85 years | 3 | 1 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 30 | 65
  Male | 23 | 28 | 13 | 64
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 33 | 32 | 32 | 97
  Asian | 9 | 10 | 10 | 29
  Other | 1 | 1 | 1 | 3
Body mass index [Median (Full Range); unit: kg/m2] | 25.9 [18.4 to 36.4] | 25.2 [17.4 to 33.0] | 24.9 [17.9 to 39.4] | 25.4 [17.4 to 39.4]

OUTCOME MEASURES:

1. Primary Outcome: Dose-response in Change in Weekly Mean of the 24-hour Average Pain Score, Using an 11-point Numeric Rating Scale (NRS), From Baseline to Week 12
Description: Since the 300 mg b.i.d. dose of EMA401 could not be initiated in the study due to premature study termination, the dose-response characterization was not performed. Specifically, only the trend test deduced from the set of candidate models was performed but the dose response estimation was not conducted.
Time Frame: Baseline up to Week 12
Population: Due to premature study termination 300 mg BID dose was not initiated
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change in Weekly Mean 24-hour Average Pain Score Using the 11 Point Numerical Rating Scale (NRS) From Baseline to Week 12
Description: The NRS is an 11-point scale ranging from zero ("no pain") to ten ("pain as bad as you can imagine") for self-reporting of pain by patients. The following parameters were evaluated using the 11-point NRS: 24-hour Average Pain Score and 24-hour Worst Pain Score Patients evaluated their "average pain" and "worst pain" during the past 24 hours in the evening prior to sleep by touching the appropriate corresponding number between zero and ten on a eDiary device.
Time Frame: Baseline up to Week 12
Population: number of patients with observed change from baseline on respective visit.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 43 | 43 | 43
scores on a scale
  Week 4 | -0.4 (0.23) | -0.9 (0.25) | -0.5 (0.23)
  Week 8 | -1.0 (0.29) | -1.0 (0.29) | -0.7 (0.30)
  Week 12 | -0.9 (0.40) | -1.2 (0.38) | -0.7 (0.40)
Statistical Analysis 1: Comparison: EMA401 25mg BID DB vs Placebo BID DB; Test type: Superiority; p = 0.689, ANCOVA; Multiplicity adjustment for the pairwise comparisons has been performed using the Hochberg procedure. Adjusted p-value 0.689; least squares mean = -0.2, 95% CI 2-sided [-1.3 to 0.9], Standard Error of Mean 0.56
Statistical Analysis 2: Comparison: EMA401 100mg BID DB vs Placebo BID DB; Test type: Superiority; p = 0.350, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean = -0.5, 95% CI 2-sided [-1.6 to 0.6], Standard Error of Mean 0.54

3. Secondary Outcome: Change in Brief Pain Inventory-Short Form Interference (BPI-SF) Mean Total Score From Baseline to Week 12
Description: The BPI-SF is a validated, self-administered (at clinic) questionnaire that assesses pain severity and its mpact on daily functions. Patients were asked to complete the 7-item pain interference scale that assessed the degree to which pain interfered with walking and other physical activity, work, mood, relations with others and sleep using a zero to ten numeric rating scale (NRS) with zero being "does not interfere" and ten being "completely interferes". A reduction in mean indicates improvement
Time Frame: Baseline up to Week 12
Measure: Mean (Standard Deviation); unit: scores on a numeric rating scale
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 43 | 43 | 43
scores on a numeric rating scale | -8.24 (12.994) | -15.03 (13.280) | -14.07 (12.535)

4. Secondary Outcome: Change in Weekly Mean of the 24-hour Worst Pain Score, Using an 11-point NRS, From Baseline to Week 12
Description: as for outcome 2
Time Frame: Baseline up to Week 12
Measure: Mean (Standard Deviation); unit: scores on numeric rating scale
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 43 | 43 | 43
scores on numeric rating scale | -1.04 (1.851) | -1.96 (2,365) | -1.49 (2.215)

5. Secondary Outcome: Number of Participants Per Patient Global Impression of Change Category at Week 12
Description: The Patient Global Impression of Change (PGIC) is a patient-reported instrument that measures change in overall status on a scale ranging from one ("very much improved") to seven ("very much worse"). The PGIC is based on the validated Clinical Global Impression of Change scale. The PGIC was to be completed by patients using the electronic tablet at the site
Time Frame: Baseline up to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 43 | 43 | 43
Participants
  Very much improved | 1 | 0 | 2
  Much improved | 2 | 5 | 7
  Minimally improved | 9 | 12 | 9
  No change | 20 | 18 | 12
  Minimally worse | 3 | 2 | 1
  Much worse | 1 | 0 | 3
  Very much worse | 0 | 0 | 0
  Missing | 7 | 6 | 9

6. Secondary Outcome: Percentage of Patients Achieving at Least 30% Pain Reduction at Week 12 on NRS 11 Point Scale
Description: The NRS is an 11-point scale ranging from zero ("no pain") to ten ("pain as bad as you can imagine") for self-reporting of pain by patients. The number of patients with observed response, i.e. a decrease of 30% /50% units in weekly mean of the 24-hour average pain score NRS. Logistic regression model with region, treatment, sex, use of PHN medications (yes/no) as factors and age and baseline NRS as covariates. An odds ratio >1 = higher chance of a clinically important improvement.
Time Frame: Baseline up to Week 12
Population: Full analysis set
Measure: Number; unit: % of participants - model adjusted rate
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 43 | 43 | 43
% of participants - model adjusted rate
  Week 4 - at least 30% pain reduction | 7.5 | 15.6 | 12.6
  Week 12 - at least 30% pain reduction | 22.3 | 29.6 | 23.6
Statistical Analysis 1: Comparison: EMA401 25mg BID DB vs Placebo BID DB; Test type: Superiority; p = 0.908, Regression, Logistic; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.3 to 3.2]
Statistical Analysis 2: Comparison: EMA401 100mg BID DB vs Placebo BID DB; Test type: Superiority; p = 0.609, Regression, Logistic; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.4 to 4.5]

7. Secondary Outcome: Percentage of Patients Achieving at Least 50% Pain Reduction at Week 12 on NRS 11 Point Scale
Description: The NRS is an 11-point scale ranging from zero ("no pain") to ten ("pain as bad as you can imagine") for self-reporting of pain by patients. The number of patients with observed response, i.e. a decrease of 50% units in weekly mean of the 24-hour average pain score NRS. Logistic regression model with region, treatment, sex, use of PHN medications (yes/no) as factors and age and baseline NRS as covariates. An odds ratio >1 = higher chance of a clinically important improvement.
Time Frame: Baseline up to Week 12
Population: Full analysis set
Measure: Number; unit: % of participants - model adjusted rate
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 43 | 43 | 43
% of participants - model adjusted rate | 12.0 | 13.4 | 10.3
Statistical Analysis 1: Comparison: EMA401 25mg BID DB vs Placebo BID DB; Test type: Superiority; p = 0.800, Regression, Logistic; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.3 to 3.2]
Statistical Analysis 2: Comparison: EMA401 100mg BID DB vs Placebo BID DB; Test type: Superiority; p = 0.653, Regression, Logistic; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.4 to 4.5]

8. Secondary Outcome: Mean Change in Insomnia Severity Index (ISI) From Baseline to Week 12
Description: Patients were asked to complete the ISI using five-point Likert-style scale as a measure of perceived sleep difficulties. Scores ranged from zero to 28, with a cut-off score of eight suggesting the presence of sub-threshold insomnia. The questionnaire assessed the severity of insomnia, satisfaction with current sleep pattern, sleep interference, "noticeability" of sleeping problem to others and concern about sleeping problems.
Time Frame: Baseline up to Week 12
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 43 | 43 | 43
scores on a scale | -1.29 (4.529) | -4.14 (5.146) | -3.44 (4.228)

9. Secondary Outcome: Change in Neuropathic Pain Symptom Inventory (NPSI) From Baseline to Week 12
Description: The Neuropathic Pain Symptom Inventory (NPSI) is a 12 item patient reported outcome measure that contains 10 descriptors representing 5 dimensions of pain (burning pain, deep/pressing pain, paroxysmal pain, evoked pain and paraesthesia/dysesthesia) and 2 temporal items designed to assess pain duration and the number of pain paroxysms. The sum of the responses to the 10 questions (all except temporal questions) was regarded as the total score and was divided by 10 (10 questions). The range of the total score and of the 5 dimensional scores is 0 to 10. Lower values represent better outcomes.
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB | Placebo BID DB
Number analyzed (Participants) | 43 | 43 | 43
scores on a scale | -0.4 (0.35) | -1.0 (0.37) | -1.0 (0.38)
Statistical Analysis 1: Comparison: EMA401 25mg BID DB vs Placebo BID DB; Test type: Superiority; p = 0.225, ANCOVA; LS mean difference = 0.6, 95% CI 2-sided [-0.4 to 1.6], Standard Error of Mean 0.49
Statistical Analysis 2: Comparison: EMA401 100mg BID DB vs Placebo BID DB; Test type: Superiority; p = 0.914, ANCOVA; LS mean difference = 0.1, 95% CI 2-sided [-1.0 to 1.1], Standard Error of Mean 0.53

10. Secondary Outcome: Plasma Pharmacokinetics (PK) Concentrations at Week 8 and 12
Description: Due to the premature termination of the study, the number of patients and observations providing PK data was much smaller than planned, and no PK model was developed. As a consequence, no PK parameters (Cmax, Tmax, AUC) were derived for this study. Only, summary statistics of the plasma concentrations were calculated
Time Frame: Week 8, Week 12
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB
Number analyzed (Participants) | 28 | 31
ng/mL
  Week 8 Prior dose n=26,31: number analyzed (Participants) | 26 | 31
  Week 8 Prior dose n=26,31 | 4.8 (86.3) | 15.9 (134.0)
  Week 8 1-3 hours n=26,31: number analyzed (Participants) | 26 | 31
  Week 8 1-3 hours n=26,31 | 75.9 (159.9) | 226.9 (138.5)
  Week 8 4-6 hours n= n=28,31 | 12.6 (86.6) | 48.9 (79.1)
  Week 12 Prior dose n=25,28: number analyzed (Participants) | 25 | 28
  Week 12 Prior dose n=25,28 | 4.9 (69.3) | 13.6 (67.7)
  Week 12 1-3 hours n=25,27: number analyzed (Participants) | 25 | 27
  Week 12 1-3 hours n=25,27 | 69.3 (163.7) | 184.00 (178.4)
  Week 12 4-6 hours n=25,28: number analyzed (Participants) | 25 | 28
  Week 12 4-6 hours n=25,28 | 13.7 (112.2) | 63.6 (98.1)

11. Secondary Outcome: Exposure-response (Decrease in Pain Intensity) Via Evaluation of Effect of EMA401 Exposure on Efficacy Variables (e.g. Change From Baseline of Pain Score), Via Descriptive Pharmacokinetics/ Pharmacodynamics (PK/PD)
Description: Due to the premature termination of the study, the number of patients providing data for PKPD analysis data was much smaller than planned and no model to correlate drug exposure (PK) with the change in the pain score (PD) was developed
Time Frame: Baseline, Week 8, Week 12
Population: Analysis was not performed
Arm/Group | EMA401 25mg BID DB | EMA401 100mg BID DB
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Treatment Emergent Adverse Events During Urgent Safety Measure (USM) Follow-Up
Description: Participants were instructed to stop taking drug immediately upon termination of study and asked to come in for two unscheduled visits for follow up safety assessments
Time Frame: Approximately from 3 weeks after end of study up to 16 weeks
Population: The Overall Number of Participants Analyzed reflects the Safety population, regardless of whether they completed the study
Measure: Count of Participants; unit: Participants
Groups:
- EMA401 25mg BID -> EMA401 25mg BID; EMA401 25mg BID -> Placebo BID: Participants on EMA401 25mg were randomized 1:1 to EMA401 25mg or placebo at end of treatment period (week 12)
- EMA401 100mg BID -> EMA401 100mg BID; EMA401 100mg BID -> Placebo BID: Participants on EMA401 100mg were randomized 1:1 to EMA401 100mg or placebo at end of treatment period (week 12)
- Placebo BID -> Placebo BID: Participants on placebo remained on placebo at end of treatment period (week 12)
Arm/Group | EMA401 25mg BID -> EMA401 25mg BID | EMA401 25mg BID -> Placebo BID | EMA401 100mg BID -> EMA401 100mg BID | EMA401 100mg BID -> Placebo BID | Placebo BID -> Placebo BID
Number analyzed (Participants) | 22 | 21 | 22 | 21 | 43
Participants
  Blood creatinine increased | 0 | 1 | 0 | 0 | 0
  Blood potassium increased | 0 | 1 | 0 | 0 | 0
  Glomerular filtration rate decreased | 0 | 1 | 0 | 1 | 0
  Alanine aminotransferase increased | 0 | 0 | 0 | 1 | 0
  Blood creatine phosphokinase increased | 0 | 0 | 0 | 1 | 0
  Blood glucose increased | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 21 days post treatment, up to maximum duration of 116 days
Description: Any sign or symptom that occurs during the study treatment plus the 21 days post treatment
Groups:
- EMA401 25 mg b.i.d.: EMA401 25 mg b.i.d.
- EMA401 100 mg b.i.d.: EMA401 100 mg b.i.d.
- Placebo b.i.d.: Placebo b.i.d.
- EMA401 25 mg b.i.d. - EMA401 25 mg b.i.d.: EMA401 25 mg b.i.d. - EMA401 25 mg b.i.d.
- EMA401 25 mg b.i.d. - Placebo b.i.d.: EMA401 25 mg b.i.d. - Placebo b.i.d.
- EMA401 100 mg b.i.d. - EMA401 100 mg b.i.d.: EMA401 100 mg b.i.d. - EMA401 100 mg b.i.d.
- EMA401 100 mg b.i.d. - Placebo b.i.d.: EMA401 100 mg b.i.d. - Placebo b.i.d.
- Placebo b.i.d. - Placebo b.i.d.: Placebo b.i.d. - Placebo b.i.d.
Arm/Group | EMA401 25 mg b.i.d. | EMA401 100 mg b.i.d. | Placebo b.i.d. | EMA401 25 mg b.i.d. - EMA401 25 mg b.i.d. | EMA401 25 mg b.i.d. - Placebo b.i.d. | EMA401 100 mg b.i.d. - EMA401 100 mg b.i.d. | EMA401 100 mg b.i.d. - Placebo b.i.d. | Placebo b.i.d. - Placebo b.i.d.
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 0/43 | 0/13 | 0/13 | 0/15 | 0/13 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/43 | 3/43 | 3/43 | 1/13 | 0/13 | 0/15 | 0/13 | 0/26
Other Adverse Events (participants affected / at risk) | 8/43 | 12/43 | 14/43 | 0/13 | 1/13 | 2/15 | 1/13 | 1/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EMA401 25 mg b.i.d. (N=43) | EMA401 100 mg b.i.d. (N=43) | Placebo b.i.d. (N=43) | EMA401 25 mg b.i.d. - EMA401 25 mg b.i.d. (N=13) | EMA401 25 mg b.i.d. - Placebo b.i.d. (N=13) | EMA401 100 mg b.i.d. - EMA401 100 mg b.i.d. (N=15) | EMA401 100 mg b.i.d. - Placebo b.i.d. (N=13) | Placebo b.i.d. - Placebo b.i.d. (N=26)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EMA401 25 mg b.i.d. (N=43) | EMA401 100 mg b.i.d. (N=43) | Placebo b.i.d. (N=43) | EMA401 25 mg b.i.d. - EMA401 25 mg b.i.d. (N=13) | EMA401 25 mg b.i.d. - Placebo b.i.d. (N=13) | EMA401 100 mg b.i.d. - EMA401 100 mg b.i.d. (N=15) | EMA401 100 mg b.i.d. - Placebo b.i.d. (N=13) | Placebo b.i.d. - Placebo b.i.d. (N=26)
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 4 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT03094195/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT03094195/SAP_001.pdf